CLINICAL TRIAL: NCT04743986
Title: The Effect of Platelet Rich Plasma on Partial Thickness Rotator Cuff Tears: A Randomized Controlled Trial
Acronym: PRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Ian King Yeung Lo, MD, FRCSC, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB14-0570
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff Injuries
Keywords: corticosteroid; platelet rich plasma; tendinopathy; partial thickness tear
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Two arm parallel randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, assessors, and the PI were blinded to the assigned treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Platelet Rich Plasma (PRP) (Experimental): Patients had 10ml venous blood drawn. Injection was performed under ultrasound guidance by one of two musculoskeletal radiologists. Injection was 3-5ml at the site of tendon pathology with the remainder of the PRP preparation infiltrated into the subacromial space. A leukocyte-poor preparation was used from a pre-packaged kit (RegenLab, Lausanne, Switzerland). The samples were centrifuged at 1500g for 5 mins to yield approx 5.5ml of 80% platelets at 1.6x concentration. The supernatant was then resuspended by inverting the tube several times and was drawn into a separate 5-ml syringe for subacromial injection.
  Interventions: Biological: Platelet Rich Plasma (PRP)
- Corticosteroid (CS) (Active Comparator): Patients had 10ml venous blood drawn. Injection was performed under ultrasound guidance by one of two musculoskeletal radiologists. The blood sample was kept for a similar time delay for centrifugation prior to injection, and was then discarded. 1ml of 40-mg/ml triamcinolone was suspended in 2ml of 0.5% bupivicaine. Injection was performed through a lateral subacromial approach after needle fenestration of the supraspinatus tendon under ultrasound visualization. CS was infiltrated into the subacromial bursa and not the tendon itself.
  Interventions: Drug: Corticosteroid (CS)

INTERVENTIONS:
Biological: Platelet Rich Plasma (PRP) — RegenLab, Lausanne, Switzerland
  Arms: Platelet Rich Plasma (PRP)
Drug: Corticosteroid (CS) — 40mg/ml triamcinolone in 2 ml 0.5% bupivicaine
  Arms: Corticosteroid (CS)

SUMMARY:
Randomized controlled trial examining platelet rich plasma versus corticosteroid injection in partial thickness rotator cuff tears or tendinopathy.

DETAILED DESCRIPTION:
We performed a randomized controlled trial on patients with imaging-shown rotator cuff tendinopathy or partial thickness tearing. Patients were randomized to receive either platelet rich plasma or corticosteroid. Follow-up was done at 6 weeks, 3 months and 12 months following injection.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* MRI or US evidence of supraspinatus tendinopathy or partial thickness tearing
* symptomatic for minimum of 3 months
* patient has exhausted a course of adequate conservative treatment (including but not limited to home/out patient physical therapy, oral analgesics, and/or shoulder injections)

Exclusion Criteria:

* prior surgical intervention on affected shoulder
* full thickness rotator cuff tear
* concomitant ipsilateral shoulder pathology (i.e. osteoarthritis, inflammatory arthritis)
* confounding cervical neck pain or radiculopathy
* more than 3 previous CS injections
* a CS injection within 6 months of study intervention
* elite level athlete
* worker's compensation case
* litigation or secondary gain issues
* unwilling or unable to provide informed consent or complete study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | change from baseline at 6 weeks, 3 months, 12 months
  visual analog scale for pain

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons shoulder score (ASES) | change from baseline at 6 weeks, 3 months, 12 months
  ASES score
Western Ontario Rotator Cuff Index (WORC) | change from baseline at 6 weeks, 3 months, 12 months
  WORC score
"Failure" | anytime from injection out to 12 months
  1) patient request for a subsequent injection, 2) consent for surgical repair, 3) undergoing surgery
Anatomic changes | 3 months and 12 months post injection
  ultrasound evidence of progression to a full thickness tear

CONTACTS AND LOCATIONS:
Overall Officials: Ian KY Lo, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available.

REFERENCES:
- [Background] Kwong CA, Woodmass JM, Gusnowski EM, Bois AJ, Leblanc J, More KD, Lo IKY. Platelet-Rich Plasma in Patients With Partial-Thickness Rotator Cuff Tears or Tendinopathy Leads to Significantly Improved Short-Term Pain Relief and Function Compared With Corticosteroid Injection: A Double-Blind Randomized Controlled Trial. Arthroscopy. 2021 Feb;37(2):510-517. doi: 10.1016/j.arthro.2020.10.037. Epub 2020 Oct 28. PMID 33127554